CLINICAL TRIAL: NCT01818999
Title: A Phase II Trial Of Ixabepilone and Stereotactic Body Radiation Therapy (SBRT) For Patients With Triple Negative Metastatic Breast Cancer
Brief Title: Ixabepilone and SBRT For Metastatic Breast Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: low accrual
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 102012-020
Record Dates: First submitted 2013-03-06; First posted 2013-03-27 (Estimated); Last update posted 2020-08-20 (Actual); Status verified 2019-01

CONDITIONS: METASTATIC BREAST CANCER
Keywords: METASTATIC BREAST CANCER
MeSH Terms: conditions — Breast Neoplasms | interventions — ixabepilone; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- arm one (Experimental): IXABEPILONE and STEREOTACTIC BODY RADIATION THERAPY (SBRT)
  Interventions: Drug: IXABEPILONE; Radiation: STEREOTACTIC BODY RADIATION THERAPY

INTERVENTIONS:
Drug: IXABEPILONE — injection
  Other Names: Ixempra
Radiation: STEREOTACTIC BODY RADIATION THERAPY — SBRT will begin between 1 and 5 weeks after the initiation of Ixabepilone. Patients will receive one, three, or five fractions.
  Other Names: SBRT

SUMMARY:
This study is being done to find the effect of Stereotactic body radiation therapy (SBRT) in combination with Ixabepilone for women with triple negative metastatic breast cancer.

DETAILED DESCRIPTION:
Ixabepilone is a FDA approved drug for the treatment of metastatic or locally advanced breast cancer after failure of chemotherapy. SBRT is a treatment method to deliver a high dose of radiation to the target, utilizing either a single dose or a small number of treatments with a high degree of precision within the body. The combination of Ixabepilone with SBRT is not an approved treatment at this time.

ELIGIBILITY:
Inclusion Criteria:

1. Biopsy proven triple negative invasive ductal or lobular metastatic breast cancer. Tumor estrogen, progesterone, and HER2 (tested by IHC or FISH) negative disease. (ER- defined as </=1% by IHC, PR- defined as </=1% by IHC, and HER2- by IHC 1+. If HER2 result by IHC is 2+ (equivocal), the tumor must be confirmed to be HER2- by FISH.
2. Age ≥ 18 years.
3. Patients must not have started Ixabepilone treatment more than 5 weeks prior to initiation of SBRT treatment.
4. Patients can have up to 6 sites of active extracranial disease(</=3 in the liver = one site and </=3 in the lung= one site) identified by CT scan, or PET/CT, within 8 weeks prior to initiation of SBRT (up to 2 contiguous vertebral metastasis will be considered a single site of disease). Maximum number of lesions treated is deemed as feasible per the treating radiation oncologist; ie: A patient with 4 right axillary lymph nodes, L1-L2 bone metastasis, 3 lung lesions, 1 left lung lesion, 2 liver lesions, and T2-T3 bone metastasis would be defined as having 6 sites of disease. Criteria to define a lesion in any location as a metastasis requiring local treatment as one of the sites for SBRT is any lesion clinically felt to be viable; defined as enlarging on CT/MRI or having persistent FDG avidity (Either SUV>3 or increase of SUV>20% over a 6 month interval).
5. Patients with skin nodules, skin invasion, or skin ulceration are eligible, if treatment with conventional radiation (at discretion of radiation oncologist) or surgery is planned. SBRT to skin nodules is not advised because of risk of skin necrosis.
6. . Patients must have had failure of an anthracycline, a taxane and capecitabine as per FDA approved criteria.
7. Performance status of ECOG 0,1, or 2.
8. Adequate organ and marrow function as defined below:

   * leukocytes ≥ 3,000/mcL
   * absolute neutrophil count ≥ 1,500/mcL
   * platelets ≥ 100,000/mcl
   * total bilirubin within normal institutional limits
   * AST(SGOT)/ALT(SPGT) ≤ 2.5 X institutional upper limit of normal
   * creatinine within normal institutional limits
9. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

   9.1 A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:
   * Has not undergone a hysterectomy or bilateral oophorectomy; or
   * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
10. Patients who would be receiving SBRT for lung tumors who are known or must have a documented forced expiratory volume in 1 second (FEV1)>/=30%.
11. Must have a CT C/A/P, or PET/CT scan within 8 weeks of enrollment.
12. Ability to understand and the willingness to sign a written informed consent

Exclusion Criteria:

1. Patients may not be actively receiving any other investigational agents.
2. Patients with untreated brain metastasis (patients can have whole brain radiation or stereotactic radiation to brain prior to enrollment).
3. Patients with leptomeningeal disease.
4. History of allergic reactions attributed to compounds of similar chemical or biologic composition to Agent(s) used in study. Patients with a history of severe reactions to Cremephor EL or its derivatives (polyoxyethylated castor oil) are ineligible as Ixabepilone contraindicated in these patients
5. Because the tolerance dose of SBRT to the gastrointestinal tract is not established, patients with metastatic disease invading the esophagus, stomach, intestines, or mesenteric lymph nodes will not be eligible.
6. Patients with more than 6 discrete extra-cranial sites.
7. Treatment for other carcinomas within the last 5 years, except cured non-melanoma skin and treated in-situ cancers.
8. Patients must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.
9. Patients must not be on concomitant CYP3A4 inhibitors or inducers (see section 4.3).

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-08 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
The effect of SBRT in combination with Ixabepilone on median progression free survival | 5 years
  To evaluate the effect of SBRT in combination with Ixabepilone on median progression free survival. Progression free survival is defined as time from initiation of treatment to progressive disease or death

SECONDARY OUTCOMES:
In-field local control and out-of field disease progression rates | 5 years
  To describe the in-field local control and out-of field disease progression rates
Safety of SBRT in combination with Ixabepilone for patients with metastatic triple negative breast cancer after prior chemotherapy | 1 year
  Evaluate the safety of SBRT in combination with Ixabepilone for patients with metastatic triple negative breast cancer after prior chemotherapy
The duration of Ixabepilone usage and time to initiation of next line systemic agent (chemotherapy or biologic agent) | 5 year
  Evaluate the duration of Ixabepilone usage and time to initiation of next line systemic agent (chemotherapy or biologic agent)
Overall survival for patients with metastatic triple negative breast treated with SBRT in combination with Ixabepilone | 5 year
  Evaluate overall survival for patients with metastatic triple negative breast treated with SBRT in combination with Ixabepilone
Generation of an immune response to tumor cells | 1 year
  Evaluate generation of an immune response to tumor cells

CONTACTS AND LOCATIONS:
Overall Officials: Asal Rahimi, MD, Principal Investigator — University of Texas
Locations (1):
- University of Texas Southwestern, Dallas, Texas, United States